CLINICAL TRIAL: NCT00596362
Title: Neoadjuvant Treatment With Intravitreal Avastin for Large Uveal Melanomas
Brief Title: Treatment With Intravitreal Avastin for Large Uveal Melanomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-040
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Results first posted 2015-04-14 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Uveal Melanoma
Keywords: Melanoma; Eye; Avastin
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Bevacizumab

ARMS (1):
- 1 (Experimental): AVASTIN
  Interventions: Drug: AVASTIN

INTERVENTIONS:
Drug: AVASTIN — a single injection of Avastin at the outpatient clinic. This will be done as follows: the pupil in the eye being treated will be enlarged with a liquid solution. Thirty minutes later, a numbing solution and then a cleansing solution will be put in to the eye. Finally, an injection of Avastin will be given into the eye. Right after this injection, your eye will be examined by your doctor. The pressure in your eye will also be tested before and after the injection. Patients will use antibiotic drops for 5 days following the injection. Following the injection, you will have weekly examinations for four weeks in the office.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of Avastin introduced into the inside of the eyeball in causing shrinkage of the uveal melanoma (tumor of the eye). Avastin is an anti-cancer drug specially designed to shrink blood vessels within tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with large uveal melanomas who elect to undergo enucleation.
* Patients diagnosed with uveal melanomas with tumor thickness > 10 mm or basal diameter > 16 mm, as measured by ultrasound examination, funduscopic examination, or transillumination.

Exclusion Criteria:

* Cases that do not meet the above criteria for tumor size will be ineligible to participate in the study.
* Patients with history of metastatic cancer (other than melanoma).
* Patients not able to provide consent for the study.
* Patients with clinical or radiographic evidence of extraocular extension of the tumor.
* Patients with a previous history of an adverse reaction to intravitreal injection.
* Patients with a poor view of the fundus due to cataract or vitreous hemorrhage.
* Patients with intravitreal silicone oil or gas tamponade.
* Patients < 18 years of age.
* Women known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Abramson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual: 04/10/2007
  Protocol Closed to Accrual: 05/13/2008
  Primary Completion Date (if applicable) 05/13/2008
  Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | AVASTIN
Started | 1
Completed | 0
Not Completed | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | AVASTIN
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: The Response of Intravitreal Avastin in Causing a Clinically Significant Reduction in Uveal Melanoma Tumor Size (Base Height and Volume).
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response, Disappearance of all target lesions; Partial Response, >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease: neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for partial response nor sufficient increase in the sum of the longest diameter of target lesions to qualify for progressive disease
Time Frame: At conclusion of study, up to 5 days
Measure: Number; unit: participants
Arm/Group | AVASTIN
Number analyzed (Participants) | 1
participants
  Progression of Disease | 1
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0

ADVERSE EVENTS:
Arm/Group | AVASTIN
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes